CLINICAL TRIAL: NCT05841537
Title: A Prospective, Post-marketing, Non-interventional Study of RISankizumab Evaluating Real-world Clinical Effectiveness in Crohn's Disease (APPRISE)
Brief Title: An Observational Study to Assess Change in Disease Activity and Adverse Events In Adult Participants With Moderate to Severe Active Crohn's Disease (CD)
Acronym: APPRISE
Status: Active, not recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P22-920
Record Dates: First submitted 2023-04-24; First posted 2023-05-03 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; CD; Risankizumab
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Risankizumab: Participants will receive risankizumab as prescribed by their physician according to local label.

SUMMARY:
Crohn's disease (CD) is an incurable chronic inflammatory disorder of the gastrointestinal tract. This study will assess how safe and effective risankizumab is in treating moderately to severely active CD in real world. Adverse events and change in disease activity will be assessed.

Risankizumab is a drug approved for the treatment of CD. All study participants will receive risankizumab as prescribed by their study doctor in accordance with approved local label. Approximately 1000 participants will be enrolled worldwide.

Participants will receive risankizumab as prescribed by their physician according to their routine clinical practice and local label. Participants will be followed for up to 36 months.

There is expected to be no additional burden for participants in this trial. Study visits may be conducted on-site or virtually as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of Crohn's disease (CD) confirmed by clinical, endoscopic and/or histological indices.
* Participants initiating risankizumab at the clinician's discretion as part of their routine clinical care.
* Participants prescribed risankizumab in accordance with the approved local label.
* Participants able to understand and communicate with the investigator and comply with the requirements of the study.
* Participants willing and able to provide authorization to use and disclose personal health information.
* Participants willing and able to participate in the collection of patient-reported data via cloud-based mobile application using a smart device (i.e., smartphone).

Exclusion Criteria:

* Females who are pregnant or breast feeding at baseline.
* Participants with any contraindication to risankizumab.
* Participants previously exposed to risankizumab.
* Participants currently participating in an interventional clinical trial.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult participants with Crohn's disease (CD)
Sampling Method: Non-Probability Sample
Enrollment: 1019 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Clinical Remission among Participants with Clinical Response at Month 3 | At Month 12
  Clinical Remission is defined as HBI <= 4. Clinical Response is defined as HBI reduction >= 3 points. The HBI is a simplified version of the Crohn's Disease Activity Index(CDAI). The HBI consists of 5 items encompassing patient-reported (well-being, symptoms) and objective (presence of abdominal mass or complications) variables. The total HBI score is the sum of the values for each of the five items. Higher HBI scores indicate greater disease activity. Scores < 5 indicate clinical remission, 5 - 7 indicate mild disease, 8 - 16 indicate moderate disease, and 16 indicate severe disease.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (154):
- Austria (6):
  - Universitaetsklinikum St. Poelten /ID# 258828, Sankt Pölten, Lower Austria
  - Medizinische Universitaet Graz /ID# 253559, Graz, Styria
  - Medizinische Universitaet Innsbruck /ID# 253563, Innsbruck, Tyrol
  - Klinikum Wels-Grieskirchen GmbH /ID# 253558, Wels, Upper Austria
  - Krankenhaus der Barmherzigen Schwestern Wien Betriebsgesellschaft m.b.H. /ID# 258824, Vienna, Vienna
  - Medizinische Universitaet Wien /ID# 261472, Vienna, Vienna
- Canada (18):
  - University of Calgary /ID# 254511, Calgary, Alberta
  - Gastroenterology and Internal Medicine Research Institution /ID# 253319, Edmonton, Alberta
  - South Edmonton Gastroenterology Research Clinic /ID# 253160, Edmonton, Alberta
  - Six08 Gastroenterology /ID# 254513, Lethbridge, Alberta
  - Dr. Sundeep Singh, Inc /ID# 254250, Kelowna, British Columbia
  - Fraser Clinical Trials Inc /ID# 254512, New Westminster, British Columbia
  - Percuro Clinical Research, Ltd /ID# 256339, Victoria, British Columbia
  - The Moncton Hospital /ID# 252960, Moncton, New Brunswick
  - Hamilton Health Sciences - McMaster University Medical Centre /ID# 255661, Hamilton, Ontario
  - Scott Shulman Medicine Professional Corporation /ID# 252961, North Bay, Ontario
  - Physician's Clinical Research Inc. /ID# 256494, North York, Ontario
  - Toronto Immune and Digestive Health Institute Inc /ID# 253946, North York, Ontario
  - Taunton surgical centre /ID# 253812, Oshawa, Ontario
  - Toronto Digestive Disease Associates /ID# 253813, Vaughan, Ontario
  - CIUSSS de l'est de l'Ile-de-Montreal - Hopital Maisonneuve-Rosemont /ID# 253522, Montreal, Quebec
  - Royal Victoria Hospital / McGill University Health Centre /ID# 254626, Montreal, Quebec
  - Diex Recherche Québec /ID# 254016, Québec, Quebec
  - CIUSSS de l'Estrie - CHUS /ID# 254591, Sherbrooke, Quebec
- France (31):
  - Hôpital l'Archet /ID# 253097, Nice, Alpes-Maritimes
  - APHM - Hopital Nord /ID# 253364, Marseille, Bouches-du-Rhone
  - CHU de Besancon - Jean Minjoz /ID# 253098, Besançon, Doubs
  - Hopital de la Cavale Blanche /ID# 253100, Brest, Finistere
  - Centre Hospitalier de Quimper /ID# 254052, Quimper, Finistere
  - CHU NIMES - Hopital Caremeau /ID# 254060, Nîmes, Gard
  - Centre Hospitalier Universitaire de Bordeaux /ID# 253095, Pessac, Gironde
  - Hôpitaux Civils de Colmar - Hôpital Pasteur /ID# 253088, Colmar, Grand Est
  - CHU Toulouse - Hopital Rangueil /ID# 253094, Toulouse, Haute-Garonne
  - CHU Montpellier - Hopital Saint Eloi /ID# 253096, Montpellier, Herault
  - CHU Reims - Hôpital Robert Debre /ID# 253366, Reims, Marne
  - Centre Hospitalier de Dunkerque /ID# 253837, Dunkirk, Nord
  - CHRU Lille - Hopital Claude Huriez /ID# 253099, Lille, Nord
  - Hopitaux Universitaires Henri Mondor - Hopital Henri Mondor /ID# 253091, Créteil, Paris
  - AP-HP - Hopital Bicetre /ID# 253093, Le Kremlin-Bicêtre, Paris
  - CHU de Nantes, Hotel Dieu -HME /ID# 254047, Nantes, Pays de la Loire Region
  - Centre Hospitalier Universitaire de Saint Etienne - Hopital Nord /ID# 253102, St-Priest-en-Jarez, Pays de la Loire Region
  - HCL - Hopital de la Croix-Rousse /ID# 256413, Lyon, Rhone
  - HCL - Hopital Lyon Sud /ID# 253104, Pierre-Bénite, Rhone
  - CHU Amiens-Picardie Site Sud /ID# 253089, Amiens, Somme
  - CHU de CAEN - Hopital de la Cote de Nacre /ID# 253368, Caen
  - CHRU Tours - Hopital Trousseau /ID# 253369, Chambray-lès-Tours
  - Clinique de Bercy /Id# 253139, Charenton-le-Pont
  - CH Annecy Genevois - Site Annecy /ID# 253103, Epagny Metz Tessy
  - CH Haguenau /ID# 253109, Haguenau
  - Clinique Jules Verne /ID# 253939, Nantes
  - AP-HP - Hopital Saint-Antoine /ID# 254044, Paris
  - CHU de Rouen /ID# 253107, Rouen
  - Centre Hospitalier Tarbes-Lourdes /ID# 253943, Tarbes
  - Hôpital Schuman /ID# 254781, Vantoux
  - Centre Medico Chirurgical Ambroise Pare Hartmann /ID# 253358, Neuilly-sur-Seine, Île-de-France Region
- Germany (37):
  - Universitaetsklinikum Heidelberg /ID# 272329, Heidelberg, Baden-Wurttemberg
  - Praxis fuer Gastroenterologie /ID# 260994, Heidelberg, Baden-Wurttemberg
  - Medizinisches Versorgunszentrum Dachau /ID# 262592, Dachau, Bavaria
  - Universitaetsklinikum Erlangen /ID# 269946, Erlangen, Bavaria
  - Gastroenterologie Opernstrasse Private Practice - Dr. Falk & Krause & Kuhn /ID# 262895, Kassel, Hesse
  - Gastroenterologische Schwerpunktpraxis /ID# 275444, Hanover, Lower Saxony
  - Mueller/Mueller-Ziehm, Hanover /ID# 261599, Hanover, Lower Saxony
  - Gastroenterologische Gemeinschaftspraxis Minden /ID# 261148, Minden, North Rhine-Westphalia
  - Magen-Darm-Zentrum-Remscheid /ID# 260681, Remscheid, North Rhine-Westphalia
  - Klinikum Worms gGmbH /ID# 269803, Worms, Rhineland-Palatinate
  - Gemeinschaftspraxis Drs. Denger und Pfitzner /ID# 261361, Friedrichsthal, Saarland
  - Zentrum für Gastroenterologie Saar MVZ GmbH /ID# 257602, Saarbrücken, Saarland
  - Praxisgemeinschaft Jerichow Schulze /ID# 262036, Jerichow, Saxony-Anhalt
  - Praxis Jessen/Grimm /ID# 257610, Altenholz, Schleswig-Holstein
  - Praxis S. Tetzlaff /ID# 257608, Buedelsdorf, Schleswig-Holstein
  - Praxis fuer Gastroenterologie /ID# 257607, Lübeck, Schleswig-Holstein
  - Praxis Heil & Mueller /ID# 265211, Andernach
  - Praxis Dr. Schiffelholz /ID# 265218, Augsburg
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 262462, Berlin
  - MVZ fuer Gastroenterlogie am Bayerischen Platz /ID# 260995, Berlin
  - Zweite Gemeinnuutzige Krankenhaus GmbH DRK Kliniken Berlin Kopenick /ID# 262711, Berlin
  - Krankenhaus Waldfriede /ID# 262341, Berlin-Zehlendorf
  - Dr. Janschek /ID# 260993, Dresden
  - Dres. Ende / Weisflog /ID# 262038, Erfurt
  - Dres. Bauer/Doerflinger /ID# 262531, Freiburg im Breisgau
  - Dres. Behrens/Fechner/Streudel /ID# 257601, Halle
  - Städtisches Kh. Heinsberg GmbH /ID# 258671, Heinsberg
  - GSGH Gastroenterologische Studiengesellschaft Herne GbR /ID# 261122, Herne
  - MVZ Dres. Al-Kadi & Partner /ID# 260996, Iserlohn
  - Dres. Breitschwerdt/Glas/Gurtler /ID# 257612, Leipzig
  - Gastropraxis Magdeburg /ID# 261340, Magdeburg
  - Gastro.Praxis am Meerbachbogen /ID# 265900, Nienburg
  - Dres. Hundorfean/Tex /ID# 261530, Nuremberg
  - Praxisklinik Nürnberg /ID# 261682, Nuremberg
  - Praxis fuer Gastroenterologie /ID# 266305, Schwerin
  - Praxis Dr. Kempelmann /ID# 261583, Tostedt
  - Dr. Schirin-Sokhan /ID# 266003, Würselen
- Israel (4):
  - Shaare Zedek Medical Center /ID# 258738, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 258737, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 257057, Tel Aviv, Tel Aviv
  - Rabin Medical Center /ID# 257058, Petah Tikva
- Italy (8):
  - Azienda Ospedaliero Universitaria Careggi /ID# 265159, Florence, Firenze
  - IRCCS Istituto Clinico Humanitas /ID# 262991, Rozzano, Lombardy
  - IRCCS Ospedale San Raffaele /ID# 265127, Milan, Milano
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata /ID# 263918, Rome, Roma
  - A.O.U. Consorziale Policlinico di Bari /ID# 264739, Bari
  - IRCCS AOU di Bologna Policlinico Sant Orsola Malpighi /ID# 265289, Bologna
  - Azienda Ospedaliera Universitaria Gaetano Martino /ID# 263592, Messina
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico /ID# 263587, Milan
- Japan (24):
  - Nagoya University Hospital /ID# 257302, Nagoya, Aichi-ken
  - Hirosaki University Hospital /ID# 256887, Hirosaki-shi, Aomori
  - Chiba University Hospital /ID# 256721, Chiba, Chiba
  - Toho University Sakura Medical Center /ID# 256668, Sakura-shi, Chiba
  - Fukuoka University Chikushi Hospital /ID# 256113, Chikushino-shi, Fukuoka
  - Fukuoka University Hospital /ID# 256718, Fukuoka, Fukuoka
  - Asahikawa Medical University Hospital /ID# 256842, Asahikawa-shi, Hokkaido
  - Sapporo Medical University Hospital /ID# 256544, Sapporo, Hokkaido
  - Hyogo Medical University Hospital /ID# 256720, Nishinomiya-shi, Hyōgo
  - Iwate Medical University Hospital /ID# 256722, Shiwa-gun, Iwate
  - Yokohama City University Medical Center /ID# 256719, Yokohama, Kanagawa
  - University Hospital Kyoto Prefectural University of Medicine /ID# 266206, Kyoto, Kyoto
  - Tohoku University Hospital /ID# 255867, Sendai, Miyagi
  - Kansai Medical University Hospital /ID# 256548, Hirakata-shi, Osaka
  - Saga University Hospital /ID# 256726, Saga, Saga-ken
  - Shiga University of Medical Science Hospital /ID# 256549, Ōtsu, Shiga
  - Hamamatsu University Hospital /ID# 256723, Hamamatsu, Shizuoka
  - Jichi Medical University Hospital /ID# 256665, Shimotsuke-shi, Tochigi
  - Institute of Science Tokyo Hospital /ID# 256669, Bunkyo-ku, Tokyo
  - The Jikei University Hospital /ID# 255741, Minato-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital /ID# 256724, Minato-ku, Tokyo
  - Kyorin University Hospital /ID# 254076, Mitaka-shi, Tokyo
  - Keio University Hospital /ID# 257239, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University Hospital /ID# 255868, Shinjuku-ku, Tokyo
- Netherlands (3):
  - Radboudumc /ID# 266526, Nijmegen, Gelderland
  - Atrium-Orbis - Zuyderland Medisch Centrum Heerlen /ID# 268085, Heerlen, Limburg
  - Elisabeth TweeSteden Ziekenhuis /ID# 267140, Tilburg, North Brabant
- Spain (12):
  - Complejo Hospitalario Universitario de Santiago (CHUS) /ID# 261195, Santiago de Compostela, A Coruna
  - Hospital Universitari de Bellvitge /ID# 261198, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marques de Valdecilla /ID# 261196, Santander, Cantabria
  - Hospital Universitario Puerta de Hierro - Majadahonda /ID# 261201, Majadahonda, Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca /ID# 261228, El Palmar, Murcia
  - Hospital Alvaro Cunqueiro CHUVI /ID# 261224, Vigo, Pontevedra
  - Hospital Juan Ramon Jimenez /ID# 261227, Huelva
  - Hospital Universitario 12 de Octubre /ID# 261200, Madrid
  - Hospital Universitario La Paz /ID# 261199, Madrid
  - Hospital Universitario de Salamanca /ID# 261197, Salamanca
  - Hospital Universitario Virgen Macarena /ID# 261225, Seville
  - Hospital Universitario Virgen del Rocio /ID# 261202, Seville
- Switzerland (7):
  - Hôpital de La Tour /ID# 259489, Meyrin, Canton of Geneva
  - Kantonsspital St. Gallen /ID# 261931, Sankt Gallen, Canton of St. Gallen
  - Gastroentérologie Beaulieu SA /ID# 259490, Lausanne, Canton of Vaud
  - University Hospital Zurich /ID# 259491, Zurich, Canton of Zurich
  - Hirslanden Klinik /ID# 262093, Zurich, Canton of Zurich
  - Inselspital, Universitaetsspital Bern /ID# 259485, Bern
  - Berner IBD Study Group /ID# 259351, Bern
- United Arab Emirates (4):
  - Sheikh Shakhbout Medical City /ID# 276665, Abu Dhabi
  - Burjeel Day Surgery Center /ID# 259188, Abu Dhabi
  - Cleveland Clinic Abu Dhabi /ID# 261681, Abu Dhabi
  - Rashid Hospital /ID# 259264, Dubai

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P22-920